CLINICAL TRIAL: NCT01342601
Title: Evaluation of the Safety and Efficacy of Ectoin Allergy Nasal Spray and Ectoin Allergy Eye Drops in the Treatment of Seasonal Allergic Rhinitis (SAR) in Children and Adolescents: a Multicenter, Double-blind, Randomised, Placebo Controlled, Parallel Group Clinical Investigation
Brief Title: Safety and Efficacy of Ectoin Allergy Nasal Spray and Ectoin Allergy Eye Drops in the Treatment of Seasonal Allergic Rhinitis (SAR) in Children and Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bitop AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PPL-041
Record Dates: First submitted 2011-04-21; First posted 2011-04-27 (Estimated); Last update posted 2011-10-13 (Estimated); Status verified 2011-10

CONDITIONS: Seasonal Allergic Rhinitis; Seasonal Allergic Conjunctivitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ectoin products (Active Comparator)
  Interventions: Device: ect4allergy Nasal Spray (ANS01) and Eye Drops (AAT01)
- Placebo products (Placebo Comparator)
  Interventions: Device: Placebo products

INTERVENTIONS:
Device: ect4allergy Nasal Spray (ANS01) and Eye Drops (AAT01) — Comparison of ANS01 and AAT01 with placebo
  Other Names: ect4allergy
  Arms: Ectoin products
Device: Placebo products — Nasal Spray and Eye drops without Ectoin
  Arms: Placebo products

SUMMARY:
Ectoin acts on membranes by forming an Ectoin-Hydro-Complex therewith providing a protection against external agents like aeroallergens. The effects of Ectoin containing nasal spray and eye drops have already been demonstrated in several studies with adult Seasonal Allergic Rhinitis (SAR) patients and it was shown that they can effectively reduce symptoms of allergic rhinitis without resulting in any significant adverse events.

The aim of this clinical investigation is to demonstrate the safety, tolerability and efficacy of Ectoin Nasal Spray and Ectoin Eye Drops in pediatric and adolescent SAR patients. It is assumed that Ectoin containing products show an excellent safety profile and very good tolerability together with a potent efficacy in the treatment of SAR.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-17 years
* diagnosed seasonal allergic rhinitis
* general good health condition other than SAR, and free of any concomitant conditions or treatment that could interfere with clinical investigation conduct, influence the interpretation of clinical investigation observations/results, or put the patient at increased risk during the clinical investigation
* Sum of Total Nasal Score (TNSS) ≥ 6
* Sum of Total Ocular Score (TOSS) ≥ 4

Exclusion Criteria:

* - Confirmed diagnosis of acute or chronic rhinosinusitis, as determined by the investigator
* History of physical findings of nasal pathology, including nasal polyps or other clinically significant respiratory tract malformations, recent nasal biopsy, nasal trauma or surgery, atrophic rhinitis, or rhinitis medicamentosa (all within the last 60 days prior to the screening visit)
* Chronic or intermittent use of intranasal, oral, intramuscular, intravenous or ophthalmic corticosteroids
* Ocular disorder other than allergic conjunctivitis, except hyperopia and myopia and strabismus
* Upper and lower airway respiratory infection or disorder [including, but not limited to bronchitis, pneumonia, chronic sinusitis, influenza, severe acute respiratory syndrome (SARS)] within 4 weeks prior to clinical investigation start or development of a respiratory infection during the run-in period
* Start of specific immunotherapy within 1 month preceding enrolment in the clinical investigation or change in dose of immunotherapy throughout the trial
* Chronic moderate to severe asthma according to GINA criteria which is treated with inhaled corticosteroids (ICS) and additional anti-asthmatic treatment. Patients with mild co-seasonal asthma must not change their dose regimen of ICS within 4 weeks prior to the enrolment into the clinical investigation nor during the clinical investigation
* Other respiratory diseases (e.g. Chronic obstructive pulmonary disease (COPD), cystic fibrosis, alpha-1-Antitrypsin deficiency, sarcoidosis, bronchiectasis, allergic alveolitis, tuberculosis, emphysema, etc.)
* on investigators discretion

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2011-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
clinically relevant changes in vital signs | 2 weeks
Incidence of adverse events | 2 weeks
Overall assessment by the patient (Rhinoconjunctivitis Quality of Life Questionnaire (PRQLQ for children aged 5-12 years or AdolRQLQ for adolescents aged 13-17 years) | 2 weeks
Change score in TNSS at visit V3 compared to baseline (V2) separately for a.m. and p.m. measurement | 2 weeks
  Total nasal symptom score: runny nose (anterior rhinorrhea/postnasal drainage), itchy nose, nasal congestion (stuffy nose) and sneezing on a 4 point scale (0=none to 3= severe)asssessed by the patient/caregiver
Change score in TOSS at visit V3 compared to baseline (V2) separately for a.m. and p.m. measurement | 2 weeks
  Total ocular symptom score: itchy eyes, red eyes, watery eyes´on a 4 point scale (0=none to 3=severe) assessed by the patient/caregiver
Change score in non-nasal score at visit V3 compared to baseline (V2) separately for a.m. and p.m. measurement | 2 weeks
  Non-nasal score: itchy ear/palate on a 4 point scale (0=none to 3=severe)assessed by the patient/caregiver
clinical relevant changes in physical examination parameters | 2 weeks
Severity of Adverse events | 2 weeks

SECONDARY OUTCOMES:
Use of rescue medication | 2 weeks
TNSS, separately for a.m. and p.m. measurement over time | 2 weeks
TOSS over time (V2, V3), separately for a.m. and p.m. measurement over time | 2 weeks
Non-nasal score over time (V2, V3), separately for a.m. and p.m. measurement over time | 2 weeks
Symptom scores separately for a.m. and p.m. measurement over time | 2 weeks
  Symptom scores: Runny nose, itchy nose, nasal congestion, Sneezing, itchy ear, itchy eyes, red eyes, watery eyes

CONTACTS AND LOCATIONS:
Overall Officials: Albrecht Bufe, Prof. Dr. med., Principal Investigator — Experimentelle Pneumologie RUB
Locations (8):
- Germany (8):
  - Kinderarzt Bleckmann, Baunatal-Großenritte
  - Dr. med. Martina Weh, Berlin
  - Experimentelle Pneumologie RUB, Bochum
  - Kinderarztpraxis Bramsche, Bramsche
  - Dr. med. Friedrich Kaiser, Hamburg
  - Dr. Marlies Bölich, Jena
  - Dr. Ralph Maier, Tuttlingen
  - Dr.med. Dieter Schlegel und Lilli Hegai, Welzheim